CLINICAL TRIAL: NCT02354898
Title: A Phase I Study of BBI503 Monotherapy in Patients With Advanced Solid Tumors, or BBI503 Plus Sorafenib Combination Therapy in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of BBI503 in Advanced Solid Tumors, or BBI503/ Sorafenib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA101003
Record Dates: First submitted 2015-01-21; First posted 2015-02-03 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumors; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

ARMS (1):
- BBI503, BBI503 and Sorafenib (Experimental)
  Interventions: Drug: BBI503; Drug: Sorafenib

INTERVENTIONS:
Drug: BBI503
Drug: Sorafenib — Sorafenib 400mg twice daily (800mg total daily dose)

SUMMARY:
This is an open-label, multicenter, phase 1 dose escalation study of BBI503 monotherapy, or BBI503 in combination with Sorafenib. This study population is adult patients with advanced solid tumors in monotherapy, or adult patients with advanced hepatocellular carcinoma in combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* ≥ 20 years of age
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI503 dose
* Females of childbearing potential must have a negative serum pregnancy test
* Adequate organ function
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Any known symptomatic or untreated brain metastases
* Pregnant or breastfeeding
* Crohn's disease, ulcerative colitis extensive gastric and small intestine resection
* Unable or unwilling to swallow BBI503 daily
* Uncontrolled concurrent disease
* Received other investigational drugs within 4 weeks prior to first dose
* Prior treatment with BBI503

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Determine of the Maximum Tolerated Dose (MTD) of BBI503 monotherapy and in combination with Sorafenib by assessing dose-limiting toxicities (DLTs) | 36 days
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately 7 months
Pharmacokinetic profile of BBI503 | 37 days

SECONDARY OUTCOMES:
Assessment of the preliminary anti-tumor activity by performing tumor assessments approximately every 8 weeks | 6 months
  The radiologic assessments will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Progression Free Survival | Approximately 7 month
  The time the participant stays on study until progression will be measured and recorded.
Overall Survival | Approximately1 year
  Participants follow-up for overall survival will occur. Maximum follow-up time is 1 year after the initial administration of the last subject.

CONTACTS AND LOCATIONS:
Locations (1):
- 5 Sites, Chiba, Etc., Japan